CLINICAL TRIAL: NCT06623487
Title: The Application Value of 68Ga-grazytracer PET in Immunotherapy for Stage III Non-small-cell Lung Cancer: a Prospective, Observationa Trial
Brief Title: The Application Value of 68Ga-grazytracer PET in Immunotherapy for Stage III Non-small-cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024-233
Record Dates: First submitted 2024-09-19; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung; PET / CT; Neoadjuvant Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neoadjuvant immunotherapy can significantly improve the pathological complete response (pCR) and major pathological response (MPR) rates in resectable stage III non-small cell lung cancer (NSCLC), and extend the event-free survival (EFS). However, the current means for evaluating its efficacy are limited. This study aims to utilize the convenient and non-invasive 68Ga-grazytracer PET imaging to detect the aggregation of CD8+ T cells in target lesions after neoadjuvant immunotherapy for stage III NSCLC, and to assess its value in efficacy monitoring, providing valuable information for clinical treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage III NSCLC, after assessment according to clinical guidelines, require neoadjuvant immunotherapy;
2. Fully-informed written consent obtained from patients;
3. Patient ability to comply with protocol requirements;
4. Age 18-75 years;
5. Life expectancy of at least 6 months.

Exclusion Criteria:

1. Patients with serious diseases that the investigator deems unsuitable for participation in the clinical study. Such as severe cardiopulmonary insufficiency, severe bone marrow suppression, severe hepatic or renal insufficiency, etc;
2. Intestinal perforation, complete intestinal obstruction;
3. Patients with uncontrolled diabetes mellitus or a fasting blood glucose value of ≥11 mmol/L on the day of the test;
4. Pregnant women and women who are potentially pregnant, as well as nursing mothers;
5. Patients with poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients are enrolled from Department of Respiratory and Critical Care Medicine, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine in China.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Predictive performance 1 | up to the end of surgery
  Sensitivity and specificity of 68Ga-grazytracer PET in predicting pathological response.

SECONDARY OUTCOMES:
Predictive performance 2 | 3 years
  Assessing the predictive value of 68Ga-grazytracer PET for adjuvant immunotherapy efficacy after surgery, as measured by disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China